CLINICAL TRIAL: NCT00289419
Title: Postoperative Analgesia After Total Hip Arthroplasty. A Comparison of Continuous Epidural Infusion and Wound Infiltration With Intraarticular Bolus Injection.
Brief Title: Intraarticular Analgesia After Total Hip Arthroplasty, a Randomised Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Professor Kjeld Soballe, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20040199
Record Dates: First submitted 2006-02-08; First posted 2006-02-09 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: Arthroplasty, Replacement, Hip; Anesthetics, Local; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine; Ropivacaine; Ketorolac; Epinephrine

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Epidural Ropivacaine, morphine
- B (Experimental)
  Interventions: Drug: Ropivacaine, Ketorolac and Adrenaline

INTERVENTIONS:
Drug: Epidural Ropivacaine, morphine — Infusion rate 4 ml/h in 48 h Solution 200 ml Ropivacaine 2mg/ml added 1 ml morphine 10 mg/ml
  Arms: A
Drug: Ropivacaine, Ketorolac and Adrenaline — Wound infiltration: 100 ml Ropivacaine 2 mg/ml added 1 ml Ketorolac 30 mg/ml and 0,5 ml adrenaline 1 mg/ml Bolus injection: 20 ml Ropivacaine 7,5mg/ml added 1 ml Ketorolac 30 mg/ml and 0,5 ml adrenaline 1 mg/ml
  Arms: B

SUMMARY:
The purpose of this study is to determine whether wound infiltration with following single-shot bolus injection with local anesthetic and NASIDs are effective in the treatment of postoperative pain after total hip replacement compared to continuous epidural infusion.

DETAILED DESCRIPTION:
Sufficient postoperative pain relief after total hip replacement is necessary to achieve normal mobilisation and a reduction of the surgical stress response. After total hip replacement epidural treatment has proven superior, with regards to pain relief, than treatment with parenteral infusions and periphery nerve blocks. Even though epidural treatment gives excellent pain relief adverse effect as motor block, urine retention, hypotension and itching occurs regularly which delays rehabilitation.

Treatment with the administration of local anesthetic in the operating field has shown its efficiency in reducing postoperative pain with a low incidence of adverse effects after various surgical procedures.

This study compares continuous epidural infusion of ropivacaine added morphine to a new technique, where ropivacaine, ketorolac and adrenaline is used to infiltrate the tissue around the hip joint during surgery, and is injected by an intraarticular catheter 8 hours postoperative.

Data of pain scores, analgesia consumption, adverse effects and mobilisation is collected for the first 4 postoperative days.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted consecutively to primary total hip arthroplasty due to arthrosis

Exclusion Criteria:

* Patients unable to provide informed consent
* Patients with contraindications for spinal anesthesia
* Patients with known hypersensitivity towards the used drugs
* Patients with severe chronic neurogenic pain
* Patients with Rheumatoid arthritis
* Patients with a daily opioid consumption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-02; Primary Completion 2006-02 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Consumption af analgesics | 96 h

SECONDARY OUTCOMES:
Side effects | 96 h
Mobilization level | 8 h
Pain scores VAS | 96 h

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Søballe, Professor, Principal Investigator — Orthopedic Center, Aarhus University Hospital, Aarhus, Denmark
Locations (1):
- Orthopedic Center, Aarhus University Hospital, Aarhus, Aarhus, Denmark